CLINICAL TRIAL: NCT05389865
Title: An Investigation Into the Epidemiology and Surgical Intervention for Proximal Aortic Disease in Scotland
Brief Title: Proximal Aortopathy in Scotland - Epidemiology and Surgical Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Aberdeen Royal Infirmary (Other); Royal Infirmary of Edinburgh (Other); Network for Inherited Cardiac Conditions Scotland (Unknown); University of Glasgow (Other)
Responsible Party: Principal Investigator, George Gradinariu, Principal Investigator, Cardiothoracic Surgery Specialty Registrar, Golden Jubilee National Hospital
Other Study IDs: IRAS 309277
Record Dates: First submitted 2022-05-06; First posted 2022-05-25 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Aortic Diseases; Aortic Dissection; Aortic Aneurysm, Thoracic; Aortic Ectasia; Aortic Valve Insufficiency; Bicuspid Aortic Valve; Marfan Syndrome; Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome
Keywords: aortic surgery; aortic root; ascending aorta; surgical outcomes; thoracic aortopathy epidemiology
MeSH Terms: conditions — Aortic Diseases; Aortic Dissection; Aortic Aneurysm, Thoracic; Aortic Valve Insufficiency; Bicuspid Aortic Valve Disease; Marfan Syndrome; Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical cohort: Adult patients (18 years of age and above) who have had a surgical intervention on the proximal aorta in the three Scottish Cardiothoracic Surgery units based in Glasgow, Edinburgh, Aberdeen.
  Interventions: Procedure: Surgery on the proximal aorta (aortic root +/- ascending aorta)
- Non-surgical cohort: - Adult patients (18 years of age and above) who have a diagnosis of proximal aortopathy, but have not had surgical intervention (non-surgical/un-intervened proximal aortopathy). This cohort will be obtained from three sources:
  1. Scottish national radiological database based on specific imaging codes
  2. Regional genetic/inherited cardiac conditions services
  3. Public Health Scotland via specific diagnostic ICD-10 codes.
  Interventions: Other: Patients diagnosed with thoracic aortopathy but not operated upon

INTERVENTIONS:
Procedure: Surgery on the proximal aorta (aortic root +/- ascending aorta) — Surgery involving replacing, repairing or reinforcing the proximal aorta (root and ascending aorta)
  Groups: Surgical cohort
Other: Patients diagnosed with thoracic aortopathy but not operated upon — Radiological size criteria or Genetic mutations associated with aortopathies
  Groups: Non-surgical cohort

SUMMARY:
The aorta is the principal arterial vessel arising from the left heart that transfers blood to the body. Certain genetic and familial disease processes are known to weaken the aortic wall resulting in dilation and potential rupture. These aortic complications carry high mortality (>25%) and current management is orientated towards early detection and preventive treatment. Aortic dilation can also result in aortic valve dysfunction leading to heart failure. The estimated UK incidence of aortic disease per year is around 10 per 100,000 individuals, with 2000 people per year dying from aortic complications.

The 2017-2020 National Adult Cardiac Surgery Audit report identified the number of people receiving surgery for aortic dissection in Scotland is per population proportionately lower compared to England (4.6 per million per year in Scotland vs. 6.6 per million per year in England). The reasons for this are unclear but may relate to the prevalence of aortic disease or a large geographic distribution with compromised access to specialized centres.

Currently surgery is recommended when the aortic diameter exceeds a certain threshold. There are several types of effective surgical procedures, but there is still limited information on their long-term outcomes and the advantage of one procedure over another.

The aims of the project are firstly to determine the clinical outcomes of the surgical procedures that are currently employed in Scotland to treat proximal aortic disease and secondly to describe the prevalence and distribution of proximal aortic disease within the Scottish population. The project will be hosted by the Golden Jubilee Research Institute. Contemporary and retrospective data will be collected from all the Scottish Cardiothoracic Surgery units which are based in Glasgow, Edinburgh and Aberdeen.

This will be the first study to analyse surgical outcomes for ascending aortic disease in Scotland, and the first to describe the epidemiology of aortic disease within the population. It is anticipated that the results will guide current surgical practise, and provide data to inform national service provision for the management of proximal aortic disease.

DETAILED DESCRIPTION:
The study has two principal aims:

1. Determine the patient demographics, procedural types and related clinical outcomes in patients who underwent surgery of the proximal thoracic aorta in Scotland
2. Describe the epidemiology of proximal aortopathy within the Scottish population, by determining the prevalence of disease, geographic distribution and patient demographics

This study will be the first to look at outcomes from a nation-wide cohort of patients following surgery of the thoracic aorta in the UK. The investigators anticipate that results from this study will inform future aortic practice and guide decisions on intervention timing and type.

Information on the prevalence and geographic distribution of aortic disease within Scotland will guide resource allocation and service configuration to allow equity in access to treatment. By raising awareness among the medical professionals and the wider community, the study should lead to improved recognition and better outcomes for patients with aortic disease.

Data will be recorded in a contemporary and retrospective manner for two patient cohorts:

1. Surgical cohort - Adult patients who have had a surgical intervention on the proximal aorta in the three Scottish Cardiothoracic Surgery units based in Glasgow, Edinburgh, Aberdeen in the last 13 years (2008 - 2021).
2. Non-surgical cohort - Adult patients who have a diagnosis of proximal aortopathy, but have not had surgery. This cohort will be obtained from three sources:

   1. Patients with a diagnosis of thoracic aortopathy identified via National Interim Clinical Imaging Procedure (NICIP) codes sourced from the Scottish Radiology Information System (RIS) and Picture Archive and Communication System (PACS) databases.
   2. Patients with a diagnosis of thoracic aortopathy identified from regional genetic services via the Network for Inherited Cardiac Conditions Scotland.
   3. Deceased patients diagnosed with proximal thoracic aortopathy or a complication thereof (aortic dissection, aortic rupture) registered at death certification and/or post mortem accessed from Public Health Scotland using ICD-10 codes.

The three data collection sites will be the Golden Jubilee National Hospital in Glasgow, the Edinburgh Royal Infirmary and Aberdeen Royal Infirmary.

The surgical cohort sample size is expected to be around 1300 patients. The non-surgical cohort is difficult to estimate, but around 500 cases yearly are expected to be identified. The research project will be hosted by the NHS Golden Jubilee Research Department.

The principal investigator (George Gradinariu) will undertake this research project as part of an postgraduate research programme (MD degree) at the University of Glasgow under the supervision of Professor Mark Danton (Congenital Cardiac Surgeon with interest in proximal aortic surgery), Professor Alex McConnachie Professor of Biostatistics, University of Glasgow) and Professor Faisal Ahmed (Samson Gemmell Chair of Child Health, University of Glasgow)

Statistical analysis will be overseen and supervised by Professor McConnachie. Descriptive statistics will be applied. Survival data will be analysed using Kaplan-Meier. Multivariable survival and logistic regression models will be used to identify variables predicting the risk of adverse outcomes. Predictive modelling to estimate the risk of adverse outcomes based on aortic root dimension will be assessed using ROC analysis. In comparing survival by procedures propensity matching will be used to minimize confounding. Analysis will be performed using R statistical analysis software (R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Surgical cohort

Inclusion Criteria:

* all adults (>18 years of age) that underwent surgical intervention on the proximal aorta in Scotland between 2008 and 2021.

Exclusion Criteria:

* Isolated surgery on the descending thoracic aorta

Non-surgical cohort

Inclusion Criteria:

- all adult patients (>18 years of age) with a radiological, genetic or post-mortem diagnosis of thoracic aortic disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Surgical cohort (Observational cohort design)- Adult patients (18 years of age and above) who have had a surgical intervention on the proximal aorta in the three Scottish Cardiothoracic Surgery units based in Glasgow, Edinburgh, Aberdeen.
  2. Non-surgical cohort (Cross-sectional design) - Adult patients (18 years of age and above) who have a diagnosis of proximal aortopathy, but have not had surgical intervention (non-surgical/un-intervened proximal aortopathy). This cohort will be obtained from three sources:
     1. Scottish national radiological database based on specific imaging codes
     2. Regional genetic/inherited cardiac conditions services
     3. Public Health Scotland via specific diagnostic ICD-10 codes.
Sampling Method: Non-Probability Sample
Enrollment: 1662 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Early survival following surgery of the proximal aorta | In-hospital or 30 days (whichever is longer)
  In-hospital or 30 days survival following surgery of the proximal aorta
Late survival following surgery of the proximal aorta | 5 years or latest available follow-up (whichever is longer)
  Long-term survival following surgery of the proximal aorta
Patient demographics and geographic distribution of thoracic aortopathy within the Scottish population | Cross-sectional analysis (2011-2021)
  Identify the demographics (age, gender, relevant risk factors) and geographic distribution (area codes) of patients diagnosed with thoracic aortopathy within the Scottish population

SECONDARY OUTCOMES:
Cardiovascular reintervention | 1 year or latest available follow-up (whichever is longer)
  Reinterventions (surgical/endovascular) related to the aortic implant or unoperated aorta Reintervention on Aortic valve (native or prosthesis)
Specified adverse events following surgery | 1 year or latest available follow-up (whichever is longer)
  episodes of endocarditis, structural valve degeneration, thromboembolism, cerebral vascular accident, anticoagulant-related bleeding
Left ventricular ejection fraction (LVEF) following surgery | 1 year or latest available follow-up (whichever is longer)
  Long-term left ventricular ejection fraction (>50% - good, 31-50% - moderate, 21-30% - poor, 20% or less -very poor) as measured by echocardiography or cardiac MRI after surgery
Aortic valve mean gradient and degree of regurgitation following surgery | 1 year or latest available follow-up (whichever is longer)
  Long-term aortic valve function as assessed by mean gradient (mmHg) and degree of regurgitation (mild/moderate/severe) in operated patients assessed by echocardiography or cardiac MRI
Genotypes and phenotypes prevalent in the Scottish population | Previous 5 years
  Identify genotypes and phenotypes in the Scottish population and assess their prevalence

CONTACTS AND LOCATIONS:
Overall Officials: George Gradinariu, MD, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To apply for further studies, beyond the current research, using the existing dataset, a research proposal submitted to the GJNH Research Department will be required. This will follow the established internal peer-review process established by the GJNH research department. If approved, a data request form will need to be submitted to the data custodian who will release the pseudo- anonymised data to the research applicant. If there is no request to extend the study then this data will be deleted.